CLINICAL TRIAL: NCT06469645
Title: The Role of Sodium Glucose Cotransporter 2 Inhibitors in the Management of Patients With Aortic Stenosis
Brief Title: The Role of SGLT2i in Management of Moderate AS
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R212199
Record Dates: First submitted 2024-06-05; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Moderate Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Valvular Heart Disease; Myocardial Fibrosis; Empagliflozin; Echocardiography; Cardiac Magnetic Resonance Scan; Cardio-pulmonary Exercise Test; Sodium Glucose Cotransporter 2 Inhibitors
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Parallel-group prospective randomised open-label blinded endpoint (PROBE) controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomised in this group will be taking the SLGT2 inhibitor (empagliflozin) on top of their regular medications for 6 months.
  Interventions: Drug: Empagliflozin 10 MG
- Control Group (No Intervention): Patients randomised in this group will continue to have their guideline directed conservative management with no changes in their regular medications.

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Participants allocated in the Intervention Group will be taking empagliflozin 10mg once a day on top of their regular medications.
  Arms: Intervention Group

SUMMARY:
Background:

The aortic valve is like a door in the heart that lets blood flow out to the body. Over time, this valve can get worn out and become too narrow, leading to a condition called aortic stenosis. When this happens, the heart has to work extra hard to push blood through the narrow valve to supply the body with what it needs. This extra effort can cause the heart muscle to become abnormally thick or to have fibrosis. For people with aortic stenosis, this can lead to more problems like feeling out of breath, chest pain, and even needing to go to the hospital. It also increases the risk of dying from heart issues. There is a type of medication called Sodium Glucose Cotransporter 2 (SGLT2) inhibitors, which has been studied in people with weak heart muscle. These medicines were found to help the heart work better and improve the pumping of blood around the body. This can be promising for patients with aortic stenosis because it might make the heart muscle stronger and protect it from damage.

Aim of research study:

The aim of this study is to investigate whether the use of the drug empagliflozin, an SGLT2 inhibitor, prevents the formation of fibrosis or the abnormal thickening of the heart muscle in patients with aortic stenosis. Using advanced imaging techniques (such as echocardiography and cardiovascular magnetic resonance), we intend to study their effect on the heart muscle of patients with aortic stenosis.

Study design:

Patients with moderate aortic stenosis will be invited for participation. Eligible consenting patients will have a baseline assessment with cardiac MRI scan, echocardiography, cardiopulmonary exercise test and validated quality of life questionnaires. They will then be randomised to receive either the SGLT2i for 6 months, or standard of care. All patients will undergo the same tests at 6 months. This way, we aim to investigate the potential changes in the heart muscle and whether the SGLT2 inhibitor prevents fibrosis or hypertrophy.

DETAILED DESCRIPTION:
Background:

Aortic stenosis represents one of the commonest valvular heart diseases in the Western World. Studies have shown that as the valvular narrowing progresses, pathological left ventricular (LV) hypertrophy and fibrosis develop. This maladaptive left ventricular remodelling is associated with adverse events and worse long-term prognosis. Currently, there is no available medication to slow down or prevent these pathological processes occurring in aortic stenosis. Evidence from recent large randomised controlled trials have demonstrated that SGLT2 inhibitors have a significant positive impact on quality of life and cardiovascular outcomes of patients with heart failure. This is a result of complex mechanisms such as attenuation of cardiac myofibroblast activity and collagen remodelling. These could be proved to be very beneficial for patients with aortic stenosis since the left ventricular pathological changes occurring in aortic stenosis share similar pathways and mechanisms with heart failure.

Study aims and objectives:

The aims of this study are to assess if:

* SGLT2 inhibitors can prevent or decelerate adverse myocardial remodelling and fibrosis.
* SGLT2 inhibitors can improve the exercise tolerance and functional capacity of patients with aortic stenosis.

Methods:

Given that the use of SGLT2 inhibitors in aortic stenosis has not been investigated before, we aim to investigate the hypotheses with an early stage randomised controlled trial. For this, patients with moderate aortic stenosis identified in the outpatient cardiology clinic will be invited to participate. Management of moderate aortic stenosis is conservative with a 'watchful waiting' approach. The participants will be randomised either to usual conservative management or to the intervention group (use of SGLT2 inhibitor on top of regular medications). They will be assessed at baseline and at 6-months following initiation of the medication. Both appointments will include evaluation of symptoms (with the use of validated questionnaire) and functional capacity (cardiopulmonary exercise test), electrocardiogram and blood tests. An echocardiogram, a scan performed routinely on a yearly basis for all patients with moderate aortic stenosis, will also be performed at baseline and at completion of the 6 months' follow-up period to evaluate for myocardial hypertrophy and remodelling. Additionally, a cardiopulmonary exercise test and a cardiac magnetic resonance scan will be performed in these two timepoints to assess for myocardial remodelling and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate aortic stenosis (aortic valve peak velocity ≥ 3m/s or mean gradient 20-40mmHg, or Aortic valve area 1.0-1.5cm2)
2. Age over 18 years

Exclusion Criteria:

1. Severe aortic stenosis (aortic valve peak velocity ≥ 4m/s or mean > 40mmHg or Aortic valve area < 1.0cm2) or planned cardiac surgery or likely need for surgery within 6 months.
2. Previous valve replacement
3. Severe hypertension (systolic >180mmHg or diastolic >100mmHg)
4. Acute pulmonary oedema or cardiogenic shock
5. Coexisting other valvular lesion of more than moderate severit.
6. Coexisting hypertrophic cardiomyopathy or amyloidosis with cardiac involvement
7. Any contraindications to MRI scanning including eGFR <30ml/min/1.73m2
8. Pregnancy or breast-feeding
9. Concomitant SGLT2 inhibitor therapy
10. Inability to receive SGLT2 inhibitor therapy
11. History of diabetes type 1 or 2
12. Severe peripheral vascular disease or non-healed leg ulcers
13. Severe liver disease
14. Rare hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in indexed extracellular volume (iECV) | 6 months
  The indexed extracellular volume (iECV) (expressed in ml/m2) will be assessed from the Cardiac Magnetic Resonance Scan at baseline and at 6 months follow-up

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction | 6 months
  Left ventricular ejection fraction (expressed in percentage, %) will be assessed from the Cardiac Magnetic Resonance Scan at baseline and at 6 months follow-up
Change in left ventricular diastolic function as assessed by the E/A ratio | 6 months
  Diastolic function will be assessed from the echocardiographic assessment at baseline and at 6 months follow-up
Change in indexed left ventricular mass | 6 months
  Change in indexed left ventricular mass (expressed in g/m2) will be assessed from the Cardiac Magnetic Resonance Scan at baseline and at 6 months follow-up
Change in percentage of myocardial uptake of late gadolinium enahncement (LGE) | 6 months
  The late gadolinium enhancement will be assessed visually and quantitatively (% of left ventricular mass) from the Cardiac Magnetic Resonance Scan at baseline and at 6 months follow-up
Change in cardiac markers (N-terminal pro b-type natriuretic peptide and high sensitivity troponin) | 6 months
  Participants will have their cardiac markers (N-terminal pro b-type natriuretic peptide and high sensitivity troponin) tested at baseline and at the 6-month follow-up visit.
Change in peak oxygen consumption (VO2) as assessed by Cardio-Pulmonary Exercise Test | 6 months
  Participants will undergo a Cardio-pulmonary Exercise Test at baseline and at 6-months follow-up. The peak oxygen consumption will be assessed and changes will be recorded.
Change in Quality of Life (QoL) as assessed with the Kansas City Cardiomyopathy Questionnaire | 6 months
  Participants will complete the Kansas City Cardiomyopathy Questionnaire at the baseline visit and at the 6-month follow up visit. The score of the Questionnaire scales from 0 to 100, with 0 denoting the worst and 100 the best possible status.

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios S. Vassiliou, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No